CLINICAL TRIAL: NCT05234775
Title: Cross-Over Study to Compare the Pharmacokinetics and Pharmacodynamics of LIB003 Process 1 and Process 2 Drug Product in Subjects With or Without Statin Therapy
Brief Title: Cross-Over Study to Compare the Pharmacokinetics and Pharmacodynamics of LIB003 Process 1 and Process 2 Drug Product
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LIB Therapeutics LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LIB003-014
Record Dates: First submitted 2022-01-17; First posted 2022-02-10 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: assignment to initial treatment group with cross over to alternate treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LIB003 (lerodalcibep) Process 1 (Experimental): 300 mg LIB003 Process 1 drug product administered SC
  Interventions: Drug: lerodalcibep
- LIB003 (lerodalcibep) Process 2 (Active Comparator): 300 mg LIB003 Process 2 drug product administered SC
  Interventions: Drug: lerodalcibep

INTERVENTIONS:
Drug: lerodalcibep — 300 mg of each drug given SC as single dose
  Other Names: LIB003

SUMMARY:
To compare the pharmacokinetics (PK), and pharmacodynamics (PD) of single subcutaneous (SC) doses of 300 mg LIB003 Process 1 (P1) and Process 2 (P2) drug product in subjects with or without statin therapy

DETAILED DESCRIPTION:
Comparison of the pharmacokinetics (PK), and pharmacodynamics (free PCSK9 and LDL-C) of single subcutaneous (SC) doses of 300 mg of both LIB003 drug product manufactured by Process 1 (P1) and Process 2 (P2) in subjects with or without statin therapy

ELIGIBILITY:
Inclusion Criteria:

* Provision of written and signed informed consent prior to any study-specific procedure
* LDL-C 70 mg/dL or above on stable diet alone or diet plus statin
* Weight of 40 kg (88 lb) and body mass index (BMI) between 17 and 42 kg/m2
* Females of childbearing potential must be using a highly effective form of birth control
* Male subjects will either be surgically sterile or agree, or partner agrees, to use highly effective form of birth control

Exclusion Criteria:

* Fasting triglyceride >400 mg/dL
* excluded lipid lowering medication
* severe renal impairment (eGFR <30 ml/min)
* fasting glucose >200 mg/dL plus HbA1c >9%
* hepatic transaminases >2.5 x ULN for laboratory
* History of any prior or active clinical condition or acute and/or unstable systemic disease compromising subject inclusion, at the discretion of the Investigator,
* NYHA class III-IV heart failure or last documented left ventricular EF <30%
* Any severe or clinically significant advert event, laboratory abnormality, intercurrent illness, or other medical condition which indicates to the Investigator that continued participation is not in the best interest of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
pharmacodynamics | 4 weeks
  comparison of free PCSK9 reductions from baseline between P1 and P2
Cmax pharmacokinetics | 4 weeks
  comparison of serum lerodalcibep Cmax between P1 and P2
AUC 0-last pharmacokinetics | 4 weeks
  comparison of serum lerodalcibep AUC 0-last between P1 and P2
T-Half pharmacokinetics | 4 weeks
  comparison of serum lerodalcibep T-HALF between P1 and P2

SECONDARY OUTCOMES:
comparison of LDL-C | 4 weeks
  comparison of serum LDL-C reductions from baseline to week 4 between P1 and P2

CONTACTS AND LOCATIONS:
Overall Officials: Traci A Turner, MD, Principal Investigator — Metabolic & Atherosclerosis Research Center
Locations (1):
- Metabolic & Atherosclerosis Research Center (MARC), Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No